CLINICAL TRIAL: NCT02797691
Title: Developing and Testing of Culturally Adapted Cognitive Behavior Therapy (CaCBT) for Pashto Speaking Pakistanis and Afghans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peshawar Medical College (Other)
Responsible Party: Principal Investigator, Muhammad Irfan, Head, Department of Mental Health, Psychiatry and Behavioural Sciences, Peshawar Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBT Pashtu 1
Record Dates: First submitted 2016-05-26; First posted 2016-06-13 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Depression, Anxiety
Keywords: Cognitive Behavior Therapy; Depression; Anxiety; Pashto; Pakistani; Afghan
MeSH Terms: conditions — Depression; Anxiety Disorders; Suppuration | interventions — Dosage Forms; Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CaCBT plus Treatment As Usual (Experimental): Receiving "CaCBT intervention" in addition to the Treatment as usual
  Interventions: Other: CaCBT; Other: Medication/ Psychotherapy
- Treatment As Usual (TAU) (Active Comparator): Receiving Treatment as usual
  Interventions: Other: Medication/ Psychotherapy

INTERVENTIONS:
Other: CaCBT — Culturally Adapted Cognitive Behaviour Therapy
  Arms: CaCBT plus Treatment As Usual
Other: Medication/ Psychotherapy — Medication/ Psychotherapy used as usual

SUMMARY:
CBT for common mental disorders has a strong evidence base in both the USA and the UK. There are wider cultural and linguistic differences between Non Pashtun and Pashtun population of Pakistan and Afghanistan and there is evidence from research to suggest that CBT might need some adaptations when working with clients from non-western background. This study, thus, aims to culturally adapt CBT for common mental disorders for Pashto speaking population in Pakistan and Afghanistan and to test the effectiveness of this adapted CBT through a small scale pilot study.

The study will be carried out using mixed methods; quantitative and qualitative. Qualitative part will consist of structured interview with a minimum of 10-15 patients; carers; and mental health professionals, respectively, using the interview questionnaires. The data will be analysed by systematic content and question analysis which will identify the emerging themes and categories. The data will then be reorganized into wider themes and categories and written for guidelines to culturally adapt therapy manual for common mental disorders.

Quantitative phase will be a RCT involving 40 patients (20 in each arm) to assess the effectiveness of a "CaCBT intervention" for Pashto speaking patients. All those who fulfill the diagnostic criteria of depressive episode or recurrent depressive disorder using ICD 10 RDC, are living near or can easily travel to the psychiatry departments in Peshawar, will be included in the study.

The intervention group of the RCT will receive CaCBT intervention in addition to the treatment as usual (TAU) while the control group receives TAU. The assessment will be carried out at base-line and at the end of therapy (8-12 weeks). Bradford Somatic Inventory (BSI), Hospital Anxiety and Depression Scale (HADS) and Brief Disability Questionnaire (BDQ)/ WHO DAS will be used to measure somatic symptoms, anxiety, depression and disability due to physical and psychological problems, respectively. Schwartz Outcome Scale will be used at follow up to measure the outcome.

ELIGIBILITY:
Inclusion Criteria:

* All those who fulfill the diagnostic criteria of Depressive episode (F32) or Recurrent depressive disorder (F33 except 33.4) or Anxiety disorder using ICD10 RDC and who live within travelling distance of the psychiatry department in Peshawar will be approached. Those patients, who have agreed to enter the study, will be assessed 2 weeks later, to fill in the baseline measures when they attend their first appointment. Patients will be asked to attend a further appointment at the end of study period and will be assessed again.

Exclusion Criteria:

* Excessive use of alcohol or drugs (using ICD 10 RDC for alcohol or drug abuse or dependence) significant cognitive impairment (for example learning disability or dementia) and active psychosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in score of Hospital Anxiety and Depression Scale (HADS) from baseline to end of therapy | 2 Months
  At baseline and after end of therapy [after 6 Weekly Sessions (in almost 8 weeks time)]

SECONDARY OUTCOMES:
Change in score of Bradford Somatic Inventory (BSI) from baseline to end of therapy | 2 Months
  At baseline and after end of therapy [after 6 Weekly Sessions (in almost 8 weeks time)]
Change in score of Brief Disability Questionnaire/ WHO DAS from baseline to end of therapy | 2 Months
  At baseline and after end of therapy [after 6 Weekly Sessions (in almost 8 weeks time)]

OTHER OUTCOMES:
Schwartz Outcome Scale | 2 Months
  At end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan, MCPS FCPS MS, Principal Investigator — Peshawar Medical College
Locations (1):
- PRIME Foundation/ Lady Reading Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No